CLINICAL TRIAL: NCT00124930
Title: A Randomized Double-blind, Parallel Group Study Comparing Olanzapine (Zyprexa) With Haloperidol (Novo-peridol) for the Relief of Nausea and Vomiting in Patients With Advanced Cancer
Brief Title: Study Comparing Olanzapine With Haloperidol for the Relief of Nausea and Vomiting in Patients With Advanced Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study suspended due to low enrollment
Sponsor: Alberta Health services (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18731; MCT 71119; ISRCTN58624349
Record Dates: First submitted 2005-07-27; First posted 2005-07-29 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Nausea; Neoplasms
Keywords: olanzapine; haldol; cancer; nausea; second line treatment; refractory nausea
MeSH Terms: conditions — Nausea; Neoplasms | interventions — Olanzapine; Haloperidol

INTERVENTIONS:
Drug: Olanzapine
Drug: Haldol

SUMMARY:
The purpose of this study is to compare the efficacy and safety of Haldol (haloperidol) and olanzapine in the control of chronic nausea with advanced cancer patients who have failed first line antiemetic therapy.

DETAILED DESCRIPTION:
The purpose of this study is to compare the efficacy and safety of haloperidol and olanzapine in the control of chronic nausea with advanced cancer patients who have failed first line antiemetic therapy.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Significant nausea/vomiting
* Failed maxeran and domperidone
* Underlying treatment of causes has failed
* Adequate cognitive function
* Communicates well

Exclusion Criteria:

* Partial/complete bowel obstruction
* Currently taking Haldol or olanzapine
* Has drug induced extrapyramidal symptoms
* Parkinson's disease
* Undergoing chemotherapy or radiotherapy (RT) to brain, abdomen, stomach or esophagus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Severity of nausea on days 3 and 5

CONTACTS AND LOCATIONS:
Overall Officials: Jose Pereira, Principal Investigator — Alberta Cancerboard
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada